CLINICAL TRIAL: NCT06969170
Title: A Phase 2a, Placebo-Controlled Randomized, Double-Blind Trial to Evaluate the Safety, Tolerability, and Preliminary Efficacy of Psilocybin Oral Solution in Adults With Generalized Anxiety Disorder
Brief Title: Safety, Tolerability, and Preliminary Efficacy of Psilocybin Oral Solution in Adults With Generalized Anxiety Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Diamond Therapeutics Inc. (Industry); Kingston Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Claudio Soares, Professor of Psychiatry, Queen's University; Director, Centre for Psychedelics Health and Research (CPHR), Queen's University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: DTI-02a-001; HC6-024-c282159 (Other: Health Canada)
Record Dates: First submitted 2025-04-15; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Generalized Anxiety Disorder (GAD)
Keywords: Psilocybin; Double-Blind; Psychedelic; Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Psilocybin; Pharmaceutical Preparations

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psilocybin Oral Solution (Experimental): Psilocybin 3mg Po (oral solution) once daily
  Interventions: Drug: Psilocybin (drug)
- Placebo (Sucralose oral solution) (Placebo Comparator): Sucralose PO (oral solution) once daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Psilocybin (drug) — Psilocybin 3mg Po (oral solution) administered daily for 28 days (Open-Label Run-in Phase) followed by Psilocybin 3mg Po (oral solution) OR Placebo for 28 days (Double-Blind Treatment Phase) in patients with Generalized Anxiety Disorder(GAD)
  Arms: Psilocybin Oral Solution
Other: Placebo — Sucralose 0.2% oral solution
  Arms: Placebo (Sucralose oral solution)

SUMMARY:
This Phase 2a clinical trial is designed to evaluate the safety, tolerability, and preliminary efficacy of a 3 mg dose of psilocybin oral solution for the treatment of Generalized Anxiety Disorder (GAD).

The study consists of three sequential phases: Screening Phase (up to 4 weeks), Open-label Run-in Phase (4 weeks), Double-blind Treatment Phase (4 weeks)

Screening Phase During the Screening Visit, participants will provide informed consent and undergo a comprehensive medical evaluation, including an abbreviated psychiatric assessment, to determine eligibility. To qualify, patients must have a clinician-rated Hamilton Anxiety Rating Scale (HAM-A) score ≥14. Additionally, participants must not be on regular anxiolytic treatment or must have discontinued such treatment at least 4 weeks prior to the start of the Open-label Run-in Phase.

Open-label Run-in Phase Eligible patients will proceed to the 4-week Open-label Run-in Phase. During this phase, patients will attend four weekly clinic visits, supplemented by weekly remote contacts (via phone or email).

At different timepoints during the OL Run-in Phase, participants will complete safety assessments, undergo cognitive testing and EEG and other patient reported outcomes (PROs).

Double-blind Treatment Phase Participants who demonstrate a treatment response during the Open-label Phase-defined as a ≥50% reduction in GAD-7 score from baseline-will be randomized 1:1 to receive either psilocybin oral solution or placebo at the Double-blind Baseline Visit. Patients not meeting the response criteria will undergo End-of-Treatment (ET) procedures at this visit.

At different timepoints during the DB Treatment Phase, participants will complete safety assessments, undergo cognitive testing and EEG and other patient reported outcomes (PROs).

Completion of the End of Treatment (ET) phase will be 2 weeks to further assess safety and PROs.

ELIGIBILITY:
Inclusion Criteria:

1. Must provide written informed consent prior to the initiation of any protocol-specific procedures.
2. Male and female adults, between 18 and 60 years of age, inclusive.
3. Meets DSM-V criteria for a primary diagnosis of GAD at Screening (duration of diagnosis ≥1 year, based on self-report), confirmed using the MINI.
4. Clinician-rated GAD-7 score ≥14 at Screening (Visit 1).
5. Clinician-rated HAM-A score ≥14 at Screening (Visit1).
6. Females must be non-pregnant and non-lactating and must fulfil at least one of the following:

   * Be surgically sterile for a minimum of 6 months (achieved through hysterectomy, oophorectomy, or bilateral salpingectomy; note that tubal ligation is not considered a method of permanent sterilization).
   * Post-menopausal for a minimum of 1 year (confirmed by follicle-stimulating hormone test).
   * Agree to avoid pregnancy and use a medically acceptable method of contraception with male sexual partners from at least 30 days prior to the study until 30 days after the study has ended (last study procedure).
   * Medically acceptable methods of contraception include any of the following:
   * Double-barrier methods (e.g., male condom, spermicide with diaphragm or spermicide with cervical cap)
   * Oral contraceptives; hormonal patch, implant or injection; or hormonal or non-hormonal intrauterine device. The male partner should use, at all times, a male condom with spermicide, should the female Patient choose to use any of these methods
   * Complete abstinence, should it be in line with the Patient's preferred and usual lifestyle.
7. Males who are able to father children must agree to use medically acceptable methods of contraception during the study and for 30 days after the last study drug administration. If a patient's partner should become pregnant during his participation in the study and for 30 days after he has completed his last study drug administration, the patient must inform study staff immediately. Medically acceptable methods of contraception include:

   * Using a condom with a female partner of child-bearing potential who is using oral contraceptives; hormonal patch, implant or injection; hormonal or non-hormonal intrauterine device; or diaphragm or cervical cap with spermicide
   * Complete abstinence, should it be in line with the patient's preferred and usual lifestyle.
8. Males must refrain from sperm donation from clinic admission to at least 30 days after the last dose of study drug.
9. Must be able to speak, read, and understand English sufficiently to allow completion of all study assessments.
10. Must be willing to comply with the requirements and restrictions of the study.

Exclusion Criteria:

1. Personal history of schizophrenia, bipolar affective disorder, delusional disorder, paranoid disorder, moderate or severe panic disorder, moderate or severe social anxiety disorder, schizoaffective disorder, moderate or severe obsessive-compulsive disorder, anorexia nervosa, bulimia nervosa, moderate or severe post-traumatic stress disorder (as assessed by the IES-R), moderate or severe personality disorder (Cluster B and Cluster C only), moderate or severe MDD (as assessed by the MINI and total scores on the MADRS > 19).
2. History or presence of any clinically significant cardiac, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, renal, or other disease at Screening, which, in the opinion of the investigator, would jeopardize the safety of the patient or the validity of the study results.
3. Recently initiated non-pharmacological treatment (e.g., Cognitive Behavioral Therapy, psychotherapy) with a psychologist or health care professional (i.e., <4 weeks prior to Screening). Patients who began a stable non-pharmacological treatment regimen >4 weeks prior to Screening will be permitted. Patients currently stable on treatment will not be permitted to modify or introduce new elements to their existing treatment regimen while enrolled in the study.
4. Currently taking pharmacological treatment for GAD or depressive symptoms on a daily basis as outlined in Table 2. Patients who discontinue pharmacological treatment within a minimum of 4 weeks or more of baseline will be permitted to enroll in the study. Sporadic, prn use of anxiolytics will be permitted; however, patients will be required to document all medication use prior to study enrollment (See Section 9.7).
5. Clinically significant abnormality on ECG, including a QT interval corrected for heart rate (Bazett; QTcB interval) of >440 milliseconds in males and >460 milliseconds in females.
6. History of allergies to the investigational product or excipients.
7. History of seizures, family history of seizures, history of head trauma, history of neurosurgery, or close family history of idiopathic generalized epilepsy or other congenital epilepsies.
8. Positive for hepatitis B virus surface antigen, hepatitis C virus antibody, or human immunodeficiency virus (HIV) antibody.
9. Positive urine drug screen at Screening , inclusive of cannabis use at a rate above 0.5g/day or 3g/week;

   - Abstinence commitment clause: Patients who use cannabis at below or up to the frequency/amount listed above may be allowed to participate if they are willing and able to discontinue use for the duration of the study period without experiencing withdrawal symptoms.
10. Current or history of moderate or severe drug or alcohol use disorder (excluding caffeine and nicotine) within the past 2 years, or lifetime history of participation in a drug rehabilitation program (other than treatment for smoking cessation).
11. Has used CNS drugs with perception-altering properties (e.g., ketamine, lysergic acid diethylamide [LSD], phencyclidine [PCP], 3,4 methylenedioxymethamphetamine [MDMA], mescaline, psilocybin, tryptamine derivatives, or ring-substituted amphetamines with perception-altering effects) on more than 1 occasion for therapeutic or non-therapeutic purposes (i.e., for psychoactive effects) within the past 6 months. History of single or episodic use will not be considered exclusionary.
12. History of suicidal ideation in the past 12 months or active/current suicidality, based on C-SSRS results.
13. Is currently using an investigational drug or device or has used such in the 30 days prior to receiving study drug.
14. Female patient is pregnant or breastfeeding.
15. Patient, in the investigator's opinion, is unsuitable for clinical study participation.

Criteria for Randomization into the Double-Blind Treatment Phase

1. Minimum 50% reduction in GAD-7 score from Open-Label Baseline Visit (Visit 1) to Double-Blind Baseline Visit

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-06 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of psilocybin | From Enrollment to the End of Treatment Phase at week 14
  Measured by:
  - Incidence, relationship and severity of Adverse Events (AEs), Adverse Events of Special Interest (AESIs) and Serious Adverse Events(SAEs)

SECONDARY OUTCOMES:
Changes in symptoms of anxiety from baseline | From Enrollment to the End of Treatment Phase at week 14
  Measured by:
  - Changes in Hamilton Anxiety Rating Scale (HAM-A) - with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe

CONTACTS AND LOCATIONS:
Locations (1):
- Kingston General Health Research Institute, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Double-blinded trial